CLINICAL TRIAL: NCT02566603
Title: A Phase 1b Open-Label, Dose Escalation Study of PRTX-100 in Adult Patients With Persistent/Chronic Immune Thrombocytopenia
Brief Title: PRTX-100-203 Open-Label, Dose Escalation Study in Adult Patients With ITP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enough data has been collected to allow analysis of the safety profile and risk-benefit.
Sponsor: Protalex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRTX-100-203; 2014-005626-35 (EudraCT Number)
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — Staphylococcal Protein A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRTX-100 (Experimental): Patients will be assigned to consecutive PRTX-100 interventions as they are enrolled into the study. Between three and six patients will be enrolled per intervention level. Intervention levels range from 3 to 24 micrograms of PRTX-100 per kilogram of patient weight. Patients may receive up to four weekly infusions of PRTX-100 over the study treatment period. PRTX-100 doses ≤ 500 μg will be infused intravenously over 30 minutes. PRTX-100 doses > 500 μg will be infused over 60 minutes. Patients will remain under observation for 4 hours after initiation of PRTX-100 dosing for safety management.
  Interventions: Drug: PRTX-100

INTERVENTIONS:
Drug: PRTX-100 — Four weekly infusions of PRTX-100 at a level of 3 micrograms of PRTX-100 per kilogram of patient weight, infused over 30 minutes, followed by four hours of observation after start of infusion.
  Other Names: SpA; Staphylococcal Protein A
Drug: PRTX-100 — Four weekly infusions of PRTX-100 at a level of 6 micrograms of PRTX-100 per kilogram of patient weight, infused over 30 to 60 minutes, followed by four hours of observation after start of infusion.
  Other Names: SpA; Staphylococcal Protein A
Drug: PRTX-100 — Four weekly infusions of PRTX-100 at a level of 12 micrograms of PRTX-100 per kilogram of patient weight, infused over 60 minutes, followed by four hours of observation after start of infusion.
  Other Names: SpA; Staphylococcal Protein A
Drug: PRTX-100 — Four weekly infusions of PRTX-100 at a level of 18 micrograms of PRTX-100 per kilogram of patient weight, infused over 60 minutes, followed by four hours of observation after start of infusion.
  Other Names: SpA; Staphylococcal Protein A
Drug: PRTX-100 — Four weekly infusions of PRTX-100 at a level of 24 micrograms of PRTX-100 per kilogram of patient weight, infused over 60 minutes, followed by four hours of observation after start of infusion.
  Other Names: SpA; Staphylococcal Protein A

SUMMARY:
Pre-clinical and clinical evaluations show that PRTX- 100 has biological activity that may lead to improved platelet levels where these are decreased due to immunological pathologies and that PRTX-100 has an acceptable safety profile. In vivo treatment with PRTX-100 has been shown to raise platelet counts in a mouse model of immune thrombocytopenia (ITP). The primary objective of the study is to assess the efficacy of PRTX-100 in terms of platelet response in patients with chronic/persistent ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to initiation of any study-related procedures
2. Male or female ≥ 18 years of age
3. ITP that has persisted for ≥ 3 months. ITP must be diagnosed in accordance The American Society of Hematology 2011 Evidence-based Practice Guideline for Immune Thrombocytopenia (Neunert et al. 2011) or the International Consensus Report on The Investigation and Management of Primary Immune Thrombocytopenia (Provan et al. 2010), as locally applicable.
4. Received ≥ 1 typical regimen for the treatment of ITP. Splenectomy is considered one regimen.
5. A mean platelet count of < 30,000/μL with no individual platelet count > 55,000/μL. The mean platelet count must be determined based on 2 platelet counts including one obtained within ≤ 7 days of first PRTX-100 dose and the other within ≤ 30 days of the first dose of PRTX-100.
6. If on corticosteroids, a dose of < 1 mg/kg prednisone per day or equivalent that has been stable for ≥ 21 days prior to the first dose of PRTX-100. High-dose pulse steroid therapy is NOT allowed within 14 days prior to the first dose of PRTX-100.
7. If on steroid-sparing adjunctive immunosuppression with cyclosporine, azathioprine, mycophenolate, or 6-mercaptopurine, the dose must have been stable for ≥ 30 days prior to the first dose of PRTX-100 and must be expected to remain stable through study Day 29, unless dose reduction is required due to toxicities. Treatment with other cytotoxic agents (e.g. cyclophosphamide, vincristine) are not allowed within three months prior to the first dose of PRTX- 100.
8. Any prior treatment with rituximab or any other anti-CD20 agent must have been > 6 months prior to the first dose of PRTX-100
9. If female, must not be pregnant (as indicated by screening negative pregnancy test), must not be nursing and must be one of the following:

   * Surgically sterile (bilateral tubal ligation, hysterectomy)
   * Postmenopausal with last natural menses > 24 months prior
   * Premenopausal and using an acceptable form of birth control. Acceptable forms of birth control include: hormonal contraceptives (implantable, oral, patch) used for ≥ 2 months prior to screening or double barrier methods (any combination of two of the following: intrauterine device [IUD], male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). All premenopausal females must have a negative urine or serum pregnancy test at screening and on Day 1 prior to first PRTX-100 treatment.

Exclusion Criteria:

1. Splenectomy ≤ 90 days prior to the first dose of PRTX-100
2. Exposure to TPO-RA within 2 weeks before inclusion
3. Previous treatment with rituximab within <6 months prior to the first dose of PRTX-100
4. Bleeding score ≥ 8 (Khellaf M et al. Haematologica 2005)
5. Unstable coronary artery disease or other medical condition (such as type 1 diabetes) that, in the investigator's opinion, might increase the risk to the patient
6. Evidence of active infection requiring antibiotic therapy ≤ 14 days prior to the first dose of PRTX-100
7. Myelodysplastic syndrome. If clinically significant anemia or pancytopenia exists, documentation of a bone marrow aspirate within 24 months prior to the first dose of PRTX- 100 showing no evidence of myelodysplasia is required.
8. Medical history systemic lupus erythematosus or any cause of secondary ITP
9. History of any treatment for cancer within the past two years other than basal cell or squamous cell carcinoma of the skin that has been treated with curative intent
10. Seropositive for human immunodeficiency virus (HIV)
11. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B or C (positive for hepatitis B surface antigen or positive anti-hepatitis C antibody test)
12. History suggestive of substance abuse
13. Clinically significant abnormalities in screening laboratory tests, including:

    * Absolute neutrophil count < 1.0 x109/L
    * Hemoglobin < 10 g/dL
    * Absolute lymphocyte count < 0.8 x109/L
    * Alanine transaminase (ALT) or aspartate transaminase (AST) > 2 x upper limit of normal (ULN)
    * Lactate dehydrogenase > 3 x ULN
    * Total bilirubin level >1.5 x ULN
    * Serum creatinine level > 0.14 mmol/L (1.6 mg/dL) in males or 0.12 mmol/L (1.4 mg/dL) in females
14. Treatment with IVIG ≤ 14 days prior to the first dose of PRTX-100
15. Treatment with an anti-Rh D antigen agent (e.g. WinRho®) ≤ 14 days prior to the first dose of PRTX-100
16. Use of any investigational drug ≤ 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the first dose of PRTX-100

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Toxicity Grading Criteria based on RCTC v 2.0 and CTCAE v 4.03 | 337 Days
  Adverse events from AEs, SAEs, infusion reactions, clinical laboratory tests (hematology, blood chemistry and urinalysis), vital signs, physical findings and ECGs over the course of the study. AE severity will be graded according to Toxicity Grading Criteria derived from published standards.

SECONDARY OUTCOMES:
Overall platelet response, change from baseline (Day 1) | Days 1, 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  Defined as a platelet count ≥ 30,000/μL and at least a doubling of baseline platelet count in patients with a baseline platelet count <30,000/μL in the absence of any concomitant rescue therapy.
Complete platelet response (number of patients) | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  The number of patients demonstrating a complete platelet response, defined as a platelet count ≥ 100,000/μL.
Time to platelet response (number of days) | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  The mean number of days from first PRTX-100 dose (Day 1) until platelet response.
Durability of platelet response (number of days) | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  The number of days from first documented platelet response to first platelet count below platelet response criteria.
Concomitant ITP medication use (number of subjects) | 337 Days
  The number of subjects considered non-responders based on concomitant ITP medication use by cohort and overall. ITP medications include thrombopoietin receptor agonists (TPO-RAs), steroid-sparing adjunctive immunosuppressive treatment (e.g. cyclosporine, azathioprine, mycophenolate), and any ITP rescue medications (e.g. IVIG) received during the study Screening and Treatment Periods.

CONTACTS AND LOCATIONS:
Overall Officials: William E Gannon, MD, Study Director — Protalex, Inc.
Locations (16):
- France (9):
  - Haut-Levêque Hospital, Pessac, Bordeaux
  - CH Lyon Sud, Pierre-Bénite, Lyon
  - Côte de Nacre Hospital, Caen
  - Mondor Hospital, Créteil
  - University Hospital, Dijon
  - Claude Huriez Hospital, Lille
  - CH La Timone, Marseille
  - CHU, Nantes
  - Canceropole, Toulouse
- United Kingdom (7):
  - Hammersmith Hospital, London, OHS
  - UCLH, London, UK
  - Guy's and St. Thomas Hospital, London, UK
  - St. Georges' Hospital, London, UK
  - Derriford Hospital, Plymouth, UK
  - University Hospital Southampton, Southampton, UK
  - Royal London Hospital, London